CLINICAL TRIAL: NCT04476706
Title: Managed Access Program (MAP) to Provide Access to Canakinumab Treatment of Cytokine Release Syndrome (CRS) in Patients With COVID-19-induced Pneumonia
Brief Title: Canakinumab MAP in COVID-19 Pneumonia With CRS
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CACZ885D2001M
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Cytokine Release Syndrome in COVID-19-induced Pneumonia
Keywords: canakinumab; Ilaris; ACZ885; COVID-19; coronavirus; pneumonia; CRS; cytokine release syndrome
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia; Cytokine Release Syndrome | interventions — canakinumab

INTERVENTIONS:
Drug: canakinumab — canakinumab
  Other Names: Ilaris; ACZ885

SUMMARY:
This is a global Managed Access Program (MAP) to provide access to canakinumab to patients with cytokine release syndrome resulting from COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Clinical diagnosis of SARS-CoV-2 virus by PCR, or by other approved diagnostic methodology, or, with presumptive diagnosis of COVID-19 (other respiratory causes ruled out and COVID-19 test pending);
* Hospitalized with COVID-19-induced pneumonia;
* Elevated CRP or ferritin levels;
* Body weight ≥ 40kg.

Exclusion Criteria:

* Eligible patients must not have a history of hypersensitivity to any drugs or metabolites of similar chemical classes as canakinumab;
* On the day of canakinumab treatment initiation; treatment with biologic immunomodulators or immunosuppressant drugs, including but not limited to TNF inhibitors and anti-IL-17 agents. Immunomodulators (topical or inhaled) for asthma and atopic dermatitis are permitted as are systemic low-dose corticosteroids (e.g. ≤10 mg prednisone per day);
* Use of tocilizumab within 3 weeks prior to dosing with canakinumab;
* Suspected or known active bacterial, fungal, or parasitic infection (besides COVID-19);
* Patients with significant neutropenia (ANC <1000/mm3);
* Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) prior to canakinumab dose.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult